CLINICAL TRIAL: NCT07398274
Title: The Örebro Severe Traumatic Brain Injury Registry (ÖrSBID): A Prospective Observational Cohort Study
Brief Title: The Örebro Severe Traumatic Brain Injury Registry
Acronym: ÖrSBID
Status: Not yet recruiting | Type: Observational
Sponsor: András Zoltán Buki (Other Government)
Responsible Party: Sponsor-Investigator, András Zoltán Buki, Principal Investigator, Region Orebro lan
Organization: Region Orebro lan (Other Government)
Other Study IDs: ÖrSBID-01; 2024-06537-01 (Other: Swedish Ethical Review Authority)
Record Dates: First submitted 2026-01-27; First posted 2026-02-09 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Severe Traumatic Brain Injury; Severe Brain Injury; Ischemic Stroke; Intracerebral Hemorrhage
Keywords: severe traumatic brain injury; severe brain injury; neurointensive care; neurocritical care; multimodal monitoring; biomarkers; longitudinal follow-up; multiomics
MeSH Terms: conditions — Brain Injuries, Traumatic; Brain Injuries; Ischemic Stroke; Cerebral Hemorrhage

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Biospecimen Retention: Samples With DNA — Biological sampled, including blood and cerebrospinal fluid collected as part of routine clinical care, are retained for biomarker, genetic and multi-omics analyses related to severe brain injury
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Severe Brain Injury Cohort: Adult patients with severe traumatic brain injury or other severe brain injuries requiring neurointensive or neurointermediate care at Örebro University Hospital

SUMMARY:
Traumatic brain injury and other severe brain injuries requiring neurointensive care are associated with high mortality, long-term disability and substantial societal burden. Despite advances in critical care, outcomes after severe brain injury remain difficult to predict and secondary brain injury plays a major role in determining prognosis.

The Örebro Severe Brain Injury Database (ÖrSBID) is a prospective observational registry that aims to systematically collect detailed clinical, physiological, imaging and biological data from adult patients with severe brain injury requiring care at the neurointesive care unit or neurointermediate care unit at Örebro University Hospital.

The purpose of the registry is to enable deep phenotyping of severe brain injury, improve understanding of secondary injury mechanisms, support outcome prediction and provide a platform for longitudinal follow-up and future research. No experimental interventions are performed as part of the study.

DETAILED DESCRIPTION:
The Örebro Severe Brain Injury Database (ÖrSBIB) is a prospective observational cohort study including adult patients with severe traumatic brain injury and other severe brain injuries of central nervous system origin., such as intracerebral hemorrhage or ischemic stroke, who require neurointensive or neurointermediate care at Örebro University Hospital.

Data are collected as part of routine clinical care and include demographic and clinical characteristics, injury severity, neurological assessments, multimodal neuromonitoring data, laboratory results, neuroimaging findings and details of medical and surgical interventions. Biological samples, including blood, cerebrospinal fluid and other clinically indicated specimens are collected according to approved protocols to enable biomarker and multiomics analyses.

Patients are followed lonitudinally, including up to 12 months after injury, to assess clinical outcomes, complications, healthcare utilization and long-term consequences of severe brain injury. The study does not involve any experimental treatments or study-specific interventions as patient care is exclusively based on international and national/local guidelines and protocols. All data collection is observational and conducted in accordance with approbal from the Swedish Ethical Review Authority (diary number 2024-06537-01)

ELIGIBILITY:
Inclusion Criteria:

* Age > 16 years
* Severe traumatic brain injury or other severe brain injury requiring neurointensive or neurointermediate care
* Admission to Örebro University Hospital

Exclusion Criteria:

* Age < 16 years < 90 years
* Non-survivable brain injury
* Patients not requiring neurointensive or neurointermediate care
* Declinced consent by patient or legal representative

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with severe traumatic brain injury or other severe brain injuries requiring neurointensive or neurointermediate care at Örebro University Hospital
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2026-02-08 (Estimated); Primary Completion 2028-02-08 (Estimated); Study Completion 2028-02-15 (Estimated)

PRIMARY OUTCOMES:
Functional outcome at 12 months | Up to 12 months after injury
  Functional outcome assessed up to 12 months after injury using clinical outcome measures and registry-based follow-up data

SECONDARY OUTCOMES:
All-cause mortality | From hospital admission (Day 1) through hospital discharge and at 12 months after injury
  All-cause mortality during acute hospitalization and during post-discharge follow-up
Healthcare utilization after severe brain injury | From hospital admission (Day 1) through hospital discharge and cumulative readmissions assessed up to 12 months after injury
  Healthcare utilization measured as length of intensive care unit stay, total hospital length of stay and number of hospital readmissions
Concentration of blood and cerebrospinal fluid biomarkers | Baseline (within 24 hours of injury) and during the acute hospital phase up to 7 days after injury
  Concentration of blood- and cerebrospinal fluid-based biomarkers obtained as part of clinical management in patients with severe traumatic brain injury

CONTACTS AND LOCATIONS:
Locations (1):
- Örebro University Hospital, Örebro, Örebro County, Sweden

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared outside of the research group and will be pseudonymized as per EU and Swedish General Data Protection Regulation (GDPR).